CLINICAL TRIAL: NCT02702102
Title: Imaging Inflammation in Patients With Diffuse Lewy Body Disease
Brief Title: Imaging Inflammation in Patients With Parkinson's Disease Dementia or Dementia With Lewy Bodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Patrick Lao, Assistant Professor of Neurological Sciences, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAQ0756; 2P50AG008702-26 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Lewy Body Disease; Dementia With Lewy Bodies; Parkinson's Disease Dementia
MeSH Terms: conditions — Lewy Body Disease | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 11C-PBR28 PET scans (Experimental): Participants will receive one IV injection of up to 20 millicuries of 11C-PBR28.
  Interventions: Drug: 11C-PBR28

INTERVENTIONS:
Drug: 11C-PBR28 — Up to 20 millicuries
  Other Names: Non-proprietary

SUMMARY:
This study uses a special type of scan called a positron emission tomography (PET) scan to take pictures of the brain. During the PET scan, a special dye called 11C-PBR28 is injected into the body.

11C-PBR28 sticks to parts of the brain where there is inflammation. The purpose of this study is to see if 11C-PBR28 can detect inflammation in patients with Parkinson's disease dementia or dementia with Lewy bodies.

11C-PBR28 is considered a drug by the Food and Drug Administration. 11C-PBR28 is not a treatment for any disease. Rather, 11C-PBR28 can be used to measure inflammation in the brain.

DETAILED DESCRIPTION:
This study is being done to see if 11C-PBR28 could be useful in diffuse Lewy body disease. Diffuse Lewy Body Disease refers to subjects with either Parkinson's disease dementia or dementia with Lewy bodies.

The hypothesis is that 11C-PBR28 binding will be greater in patients with diffuse Lewy body disease than in controls, with largest differences in temporal and limbic regions of the brain.

Participants will have a medical history and examination. This will include questions about thinking and memory. Participants will have blood drawn for routine lab tests. Blood will also be tested for a special genetic test to make sure the 11C-PBR28 scan will work. A special genetic blood test will also be done to see if participants have genes that are associated with dementia with Lewy bodies or other causes of dementia. Participants will not receive the results of these special genetic tests. Participants will also have a magnetic resonance imaging (MRI) scan of the brain.

If a participant still meet the inclusion and exclusion criteria after these procedures are done, then the participant will have one PET scan using 11C-PBR28. This scan will take place at the Columbia University Medical Center Kreitchman PET Center. On the day of the PET scan you will have an intravenous (IV) catheter (tube) placed in the participant's arm. The participant will also have an arterial catheter placed in an artery of your wrist. Participant will be asked to lay down on a PET scanner. A CT scan will be taken of the participant's head. A small amount of 11C-PBR28 will be injected into the IV. A member of the study team will draw blood from the arterial catheter. The PET scan will last 90 minutes. The participant will be asked to lay still during the scan.

The amount of radiation from the 11C-PBR28 PET scan is up to 20 millicuries. Similar amounts of 11C-PBR28 have been given to over 100 human subjects in prior studies.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients:

  1. Age 60 and older.
  2. Meet criteria for either a) dementia with Lewy bodies, or b) Parkinson's disease dementia.
  3. Written and oral fluency in English.
  4. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
  5. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.
* Inclusion criteria for controls:

  1. Age 60 and older.
  2. Normal cognitive and motor function based on neurological examination.
  3. Written and oral fluency in English.
  4. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
  5. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain other brain disorders.
2. Certain significant medical conditions. Examples are uncontrolled epilepsy or multiple serious injuries.
3. Contraindication to MRI scanning.
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.
6. Low affinity binding on TSPO genetic screen
7. Currently taking anticoagulant drugs (e.g., warfarin).
8. Women of childbearing potential.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kreisl, MD, Study Director — Columbia University; Patrick Lao, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 11C-PBR28 PET Scans
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 11C-PBR28 PET Scans: Elderly participants will receive one IV injection of up to 20 millicuries of 11C-PBR28.
Arm/Group | 11C-PBR28 PET Scans
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  50-59 years old | 0
  60-69 years old | 1
  70-79 years old | 3
  80-89 years old | 1
  90-99 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Absolute 11C-PBR28 Binding (Total Distribution Volume Corrected for Free Fraction in Plasma)
Description: Using Arterial blood sampling and 11C-PBR28 PET scan uptake, a Vt was found (as opposed to an SUVR) for target regions. Volume of distribution (VT) of a radioligand is defined as the ratio of the radioligand concentration in tissue target region (CT, kBq·cm-3) to that in plasma (CP, kBq·mL-1) at equilibrium.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: kBq·cm-3 / kBq·mL-1
Arm/Group | 11C-PBR28 PET Scans
Number analyzed (Participants) | 5
kBq·cm-3 / kBq·mL-1 | 0.15 (0.17)

2. Secondary Outcome: Relative 11C-PBR28 Binding
Description: Standardized Uptake Value Ratio (SUVR) measured on PET scan using 11C-PBR28.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: SUV ratio
Arm/Group | 11C-PBR28 PET Scans
Number analyzed (Participants) | 5
SUV ratio | 0.94 (0.20)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | 11C-PBR28 PET Scans
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT02702102/Prot_SAP_000.pdf